CLINICAL TRIAL: NCT03201107
Title: Effects of a Program of Pilates Exercises on Obesity, Sarcopenic, Risk of Falls and Health in Spanish Postmenopausal Women
Brief Title: Obesity, Sarcopenic, Risk of Falls in Spanish Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Physiotherapy, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UJaen
Record Dates: First submitted 2017-06-22; First posted 2017-06-28 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Fall Due to Loss of Equilibrium
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The assignment to the groups will be of simple random type and hidden. Those responsible for admitting patients to the intervention phase will not know what group has been assigned each. This assignment will be made in advance by a researcher who will not intervene in the later stages of evaluation, intervention, data recording and elaboration of database. The assignment will be communicated through sealed and totally opaque envelopes.
  All measurements given above will be made both to the control group and to the experimental group just prior to the start of the intervention, and immediately after and six months after the end of this period, and the results will be recorded in a data record
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates group (Experimental): This group receives physical training based on pilates exercises
  Interventions: Other: Pilates
- No intervention group (No Intervention): This group does not receive any treatment

INTERVENTIONS:
Other: Pilates — Training based on a basic level Pilates exercise program will be as follows:
  A duration of weeks with a frequency of 2 sessions a week and with a duration of 55 minutes each. The exercises to be performed will be divided into three distinct phases: warm-up, lasting 15 minutes; Main part with a duration of 30 minutes and the return to calm, based mostly on stretching and with a duration of 10 minutes. The repetitions of the exercises will be between 5 and 10 according to the difficulty.
  Arms: Pilates group

SUMMARY:
To analyze the effects of a Pilates exercise program on obesity, sarcopenic, risk of falls and health in Spanish postmenopausal women.

DETAILED DESCRIPTION:
This is a randomized clinical trial of single-blind with 2 arms (Control group and experimental group), in which a pre-treatment-postest design has been used.

The study will define two groups:

* A control group (CG) that will not be submitted to treatment, which will be evaluated in the pre and post phase of the study. Participants assigned to this group will receive general advice on the positive effects of regular physical activity and will be given a guide to recommendations for promoting physical activity.
* An experimental group (GE) that after an initial evaluation will undergo a physical training program based on Pilates exercises.

Once the intervention is finished, it will be submitted to a final evaluation to see if there is a difference or not with the results obtained at the beginning.

ELIGIBILITY:
Inclusion Criteria:

* No menstrual activity for at least 12 months.
* Present obesity and / or sarcopenic.
* Do not participate in a weight loss program.
* Be able to understand the instructions, programs and protocols of this project.

Exclusion Criteria:

* Contraindications for conducting physical tests.
* Diseases that limit the static and dynamic balance and physical activity. -
* Central or peripheral vestibular or nerve alterations.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 107 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Dynamometer | At the beginning and at three months
  Dynamometer will be employed to assess hand grip stregth.
ABC-16 (Activities Specific Balance Confidence Scale) | At the beginning and at three months
  Questionnaire that assesses balance confidence in performing activities of daily living.
FES-I (Falls Efficacy Scale-International) | At the beginning and at three months
  Questionnaire that evaluates the fear of falling.
Barthel index | At the beginning and at three months
  Measures disability or dependence in activities of daily living
KATZ INDEX | At the beginning and at three months
  Is a widely used tool to assess the level of independency in older adults.
FSS (Fatigue Severity Scale) | At the beginning and at three months
  A self-report scale describing the severity of fatigue and the impact of fatigue on activities of daily living.
PSQI (Pittsburgh Sleep Quality Index) | At the beginning and at three months
  A simple and valid assessment of both sleep quality and disturbance that might affect sleep quality.
HADS (The Hospital Anxiety And Depression) | At the beginning and at three months
  A reliable, valid and practical screening tool for identifying and quantifying anxiety and/or depression in non- patients.
SF-36 (The Short Form-36 Health Survey) | At the beginning and at three months
  Used extensively for assessing health-related quality of life.
MRS (Menopause Rating Scale): | At the beginning and at three months
  Assesses the severity of menopause-related complaints and the impact on health-related quality of life.
FSFI (Female Sexual Function Index) | At the beginning and at three months
  Is a brief questionnaire that evaluates sexual functioning in women.
INBODY | At the beginning and at three months
  Valid and reliable tool to quantify and measure the 4 major components of body composition: Water, Protein, Minerals and Fat.
Bone Mineral Content (BMC) | At the beginning and at three months
  Is mineral mass in bone.
Body Weight | At the beginning and at three months
  Is the sum of Body Fat and Fat Free Mass.
Skeletal Muscle Mass (kg) | At the beginning and at three months
  Is computed based on muscle mass of the limbs, which is almost composed of skeletal muscle and takes up about 70% of total body skeletal muscle
Lean Body Mass | At the beginning and at three months
  The amount of lean body mass.
Body Fat Mass | At the beginning and at three months
  The standard range of Body Fat Mass is ascertained by calculating an examinee Body Fat Mass as compared to the standard weight and standard Body Fat Mass.
Percent of Body Fat (%) | At the beginning and at three months
  Indicates the percentage of body fat to body weight.
BMI (Body Mass Index) | At the beginning and at three months
  Is calculated from the formula, Weight (kg) / Height2 (m2), whose unit is kg/m2. It is a rough indicator of total body fat.
Segmental Analysis | At the beginning and at three months
  Is the technology that assumes the body as five cylinders of four limbs and trunk and measures the impedance of these parts separately. Segmental body composition analysis provides segmental measurement of body water, muscle mass, and fat free mass.
OPTOGAIT | At the beginning and at three months
  Is an innovative system for movement analysis and functional assessment of patients with normal or pathological conditions. REACTION TEST: This test detects the time between one optical/acoustic impulse and the patient's movement. It can be used to measure simple reactions or more complex movements
TUG (Timed Up and Go test) | At the beginning and at three months
  Is a simple test used to assess a person's mobility and physical function
CT10P | At the beginning and at three months
  Test that evaluates the balance by walking along a straight line.
STABILOMETRIC PLATFORM | At the beginning and at three months
  Instrument composed of resistive pressure sensors, used to measure the static or postural balance. The test was performed under both eyes-open and eyes-closed conditions.
X mean | At the beginning and at three months
  Mean value of the lateral oscillations of the Pressure Center
Y mean | At the beginning and at three months
  Mean value of the anteroposterior oscillations of the Pressure Center
RMS X | At the beginning and at three months
  Mean position of the center of pressure in the mediolateral plane.
RMS Y | At the beginning and at three months
  Mean position of the center of pressure in the anteroposterior plane
Length | At the beginning and at three months
  Length of the path described by the center of pressure.
Area | At the beginning and at three months
  Area of the path described by the center of pressure.
Velocity | At the beginning and at three months
  Is an estimate of the average velocity of displacement of the center of pressures of the subject during the whole test.
Isaac test | At the beginning and at three months
  Questionnaire that measures verbal fluency.
trail making test part a y b | At the beginning and at three months
  Neuropsychological test of visual attention and task switching.
mmse (mini-mental state examination) | At the beginning and at three months
  A tool that can be used to systematically and thoroughly assess mental status.
chair sit and reach test | At the beginning and at three months
  To test low back and hamstring flexibility.
back scratch test | At the beginning and at three months
  To measure general shoulder range of motion.
30-second chair stand test | At the beginning and at three months
  To test leg strength and endurance.
height | At the beginning and at three months
  The distance between the lowest and highest points of a person standing upright.
waist circumference | At the beginning and at three months
  Is used to assess central fat distribution and degree of abdominal obesity.
hip circumference | At the beginning and at three months
  It is the greatest circumference of hip
waist-to-hip ratio | At the beginning and at three months
  Is the dimensionless ratio of the circumference of the waist to that of the hips. This is calculated as waist measurement divided by hip measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Center of active participation of seniors of Jaén "Catedral", Jaén, Spain

IPD SHARING:
Plan to Share IPD: No